CLINICAL TRIAL: NCT05801380
Title: Monitoring Drug Efficacy Through Multi-omics Research Initiative in Alzheimer's Disease
Brief Title: Monitoring Drug Efficacy in Patients with Alzheimer's Disease
Acronym: MEMORI-AD
Status: Recruiting | Type: Observational
Sponsor: University of the Philippines (Other)
Responsible Party: Principal Investigator, Fresthel Monica Climacosa, Associate Professor, University of the Philippines
Other Study IDs: SJREB-2022-15
Record Dates: First submitted 2023-03-10; First posted 2023-04-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease
Keywords: multiOMICs; drug response
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. 10 mL of venous blood
  2. Fecal specimen
  3. 30 mL of urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Alzheimer's disease patients with AChE inhibitor monotherapy: This cohort includes those with the disease and given AChE inhibitor monotherapy only
  Interventions: Drug: AChE inhibitor monotherapy
- Alzheimer's disease patients given AChE inhibitor and NMDA receptor anatgonist combination therapy: This cohort includes those with the disease, given AChE inhibitor and NMDA receptor antagonist combination therapy
  Interventions: Drug: AChE inhibitor and NMDA receptor antagonist combination therapy

INTERVENTIONS:
Drug: AChE inhibitor monotherapy — This is a drug treatment using Donepezil only
  Other Names: Donepezil
  Groups: Alzheimer's disease patients with AChE inhibitor monotherapy
Drug: AChE inhibitor and NMDA receptor antagonist combination therapy — This is a drug treatment combining Donepezil and Memantine
  Other Names: Donepezil and Memantine combination therapy
  Groups: Alzheimer's disease patients given AChE inhibitor and NMDA receptor anatgonist combination therapy

SUMMARY:
This study will explore the different factors associated with drug response to acetylcholinesterase (AChE) inhibitor (donepezil) and NMDA receptor antagonist (memantine) in patients with Alzheimer's Disease.

DETAILED DESCRIPTION:
These patients will be grouped according to the medications prescribed by their attending physician at baseline, 3rd month, and 6th month of follow up:

1. Alzheimer's Disease patients given AChE inhibitor monotherapy
2. Alzheimer's Disease patients given combination therapy of AChE inhibitor and NMDA receptor antagonist

They will be observed for treatment response for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed with mild or moderate dementia using the Montreal Cognitive Assessment and Clinical Dementia Rating (CDR) performed by a licensed psychometrician
* clinically diagnosed by an expert adult neurologist as having probable AD using the National Institute of Neurological and Communicative Disorders and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* treatment naive for any acetylcholinesterase inhibitors or memantine OR those who have not taken any acetylcholinesterase inhibitors or memantine in the last three months for any reasons except for adverse drug reaction
* age 65 years old
* residing in the National Capital Region
* able to read and understand written and spoken English and Filipino

Exclusion Criteria:

* with structural or vascular causes of dementia other than subcortical lacunes (2 or less) as seen in plain CT scan
* dementia diagnosis other than AD as determined by an expert adult neurologist
* with untreated depression or related psychiatric disorders in the last 6 months
* use of systemic antibotics in the previous three months prior to providing fecal specimens
* use of corticosteroids, immune stimulating medications, and immunosuppressive agents within the past 2 weeks or those who regularly need them for immune-related disorders
* use of proton-pump inhibitors, H2-receptor antagonists, H2-receptor antagonists, tricyclic antidepressants, narcotics, anticholinergic medications, laxatives or anti-diarrheal in the past 4 weeks
* large doses of commercial probiotics consumed (greater than or equal to 108 cfu or organisms per day)
* major dietary change during previous month (defined as eliminating or significantly increasing a major food group)
* major GI tract surgery in the past 5 years, with the exception of cholecystectomy and appendectomy
* major bowel resection at any time
* active uncontrolled GI disorders or diseases, including inflammatory bowel disease, indeterminate colitis, irritable bowel syndrome, persistent infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, recurrent Clostridium difficile infection, untreated Helicobacter pylori infection, chronic constipation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All elderly patients from (1) University of the Philippines - Philippine General Hospital; (2) The Medical City; and (3) Cardinal Santos Medical Center that meet the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Change in gene signatures | Baseline, 3rd month, 6th month
  Gene signatures obtained via whole exome sequencing
Change in gut microbiome metabolome signatures | Baseline, 3rd month, 6th month
  Gut microbiome signatures obtained via gut microbiome shotgun metagenomic profiling
Change in metabolome signatures | Baseline, 3rd month, 6th month
  Metabolome signatures obtained via untargeted metabolomic profiling
Change in levels of cognition using the Montreal Cognitive Assessment-Philippines (MoCA-P) | Baseline, 3rd month, 6th month
  Montreal Cognitive Assessment-Philippines (MoCA-P) is an assessment tool used to measure mild cognitive impairment and early Alzheimer's disease. Scores range from 0-30. A score below 21 signifies mild cognitive impairment or early Alzheimer's disease.
Change in levels of cognition using the Mini-Mental State Examination (MMSE) | Baseline, 3rd month, 6th month
  The Mini-Mental State Examination (MMSE) is an assessment tool used to measure cognitive aspects of mental functions, with scores ranging from 0-30, with lower scores indicating increasing levels of cognitive impairment.
Change in levels of cognition using the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) | Baseline, 3rd month, 6th month
  Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) assesses the severity of cognitive dysfunction in Alzheimer's Disease patients. Scores range from 0-94, with higher scores indicating increased levels of cognitive dysfunction.

SECONDARY OUTCOMES:
Change in levels of functioning using the Katz Index of Activities of Daily Living (IADL) scale | Baseline, 3rd month, 6th month
  The Katz IADL assesses the patient's need for assistance in performing basic activities of daily living. Possible scores range from 0-12, with a higher score indicating better levels of functioning.
Change in levels of functioning using the Lawton instrumental activities of daily living (IADL) scale | Baseline, 3rd month, 6th month
  The Lawton IADL assesses the patient's ability to carry out more complex tasks of daily living. Scores range from 0 indicating low function and dependent up to 16 indicating highly functional and independent.
Changes in levels of behaviour using the Neuropsychiatric inventory (NPI) scale | Baseline, 3rd month, 6th month
  The neuropsychiatric inventory (NPI) scale is an informant-based interview that assesses neuropsychiatric symptoms in terms of frequency, severity, and levels of distress. Scores range from 0 to 144, with higher scores indicating the presence of more neuropsychiatric symptoms.
Change in levels of family functioning using the Filipino Family APGAR | Baseline, 3rd month, 6th month
  Filipino family APGAR is a tool to assess family functioning based on five parameters: Adaptability, Partnership, Growth, Affection, and Resolve. The total scores range from 0 to 10 with higher scores indicating higher levels of satisfaction with family functioning.
Change in levels of family functioning using the SCREEM Family Resources Survey (SCREEM-RES) | Baseline, 3rd month, 6th month
  The SCREEM Family Resources Survey (SCREEM-RES) is a tool used to measure family resources that the family utilizes to cope with difficult situations. Scores range from 0 to 36, with higher scores indicating adequate levels of family resources.

CONTACTS AND LOCATIONS:
Overall Officials: Fresthel Monica M Climacosa, MD, PhD, Principal Investigator — University of the Philippines Manila; Veeda Michelle M Anlacan, MD, Principal Investigator — University of the Philippines Manila
Locations (1):
- Philippine General Hospital, Manila, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Climacosa FMM, Anlacan VMM, Gordovez FJA, Reyes JCB, Tabios IKB, Manalo RVM, Cruz JMC, Asis JLB, Razal RB, Abaca MJM, Dacasin AB, Espiritu APN, Gapaz NCLL, Lee Yu MHL. Monitoring drug Efficacy through Multi-Omics Research initiative in Alzheimer's Disease (MEMORI-AD): A protocol for a multisite exploratory prospective cohort study on the drug response-related clinical, genetic, microbial and metabolomic signatures in Filipino patients with Alzheimer's disease. BMJ Open. 2024 Nov 27;14(11):e078660. doi: 10.1136/bmjopen-2023-078660. PMID 39608999